CLINICAL TRIAL: NCT03510689
Title: Genetics and Heart Health After Cancer Therapy
Acronym: Gene-HEART
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 13117
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Hereditary Breast/Ovarian Cancer (brca1, Brca2); Heart Diseases; Drug-Induced Cardiomyopathy
Keywords: Cardio-oncology
MeSH Terms: conditions — Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome; Heart Diseases | interventions — Echocardiography; Exercise Test; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Subjects with genetic testing confirming deleterious mutations in BRCA1 or BRCA2 whose prior treatment for breast cancer includes anthracycline exposure. All groups have same schedule of study procedures, including echocardiography, cardiopulmonary exercise testing, and blood collection.
  Interventions: Diagnostic Test: echocardiography; Other: Cardiopulmonary Exercise Testing; Other: Blood Collection
- Group 2: Subjects with genetic testing confirming deleterious mutations in BRCA1 or BRCA2 whose prior treatment for breast cancer does not include anthracycline exposure. All groups have same schedule of study procedures, including echocardiography, cardiopulmonary exercise testing, and blood collection.
  Interventions: Diagnostic Test: echocardiography; Other: Cardiopulmonary Exercise Testing; Other: Blood Collection
- Group 3: Subjects with genetic testing confirming no mutation in BRCA1 or BRCA2 whose prior treatment for breast cancer includes anthracycline exposure. All groups have same schedule of study procedures, including echocardiography, cardiopulmonary exercise testing, and blood collection.
  Interventions: Diagnostic Test: echocardiography; Other: Cardiopulmonary Exercise Testing; Other: Blood Collection

INTERVENTIONS:
Diagnostic Test: echocardiography — Resting echocardiograms (Vivid E9 or E95, GE Healthcare) with conventional measures of systolic and diastolic function, in conjunction with posthoc quantitation of novel measures of strain and strain rate will be obtained at each study time point.
Other: Cardiopulmonary Exercise Testing — A cardiopulmonary exercise test (CPET, also called V02 test) will be completed at each study time point utilizing a standard clinical protocol, on either a stationary bike or treadmill. The purpose of this test is to estimate maximal oxygen consumption (V02 max) as in index of cardiopulmonary fitness. Resting ECG, heart rate, and BP will be obtained prior to beginning the test, during each stage of the test and for 5 minutes after the test is stopped.
Other: Blood Collection — We will obtain blood samples (approximately 16mL) at baseline and (approximately 12mL) at each follow-up visit. Typically these will be drawn via peripheral venipuncture, however if patients have a port-a-cath in place, blood may be drawn from the port instead.

SUMMARY:
The overall objective of this study is to use patient-centered in vitro and in vivo models to answer the fundamental question of whether or not pathogenic mutations in BRCA1/2 result in an increased risk of CV disease

ELIGIBILITY:
Inclusion Criteria

* ≥18 years of age
* Initial diagnosis of Breast Cancer in 2005 or later
* Documented BRCA testing (results from a local laboratory are acceptable) showing

  * confirmation of a germline mutation in BRCA1 or BRCA2 that is predicted or suspected to be deleterious OR
  * confirmation that no mutation was detected in BRCA1 or BRCA2
* Non-carriers will have been treated with an anthracycline-based chemotherapy regimen; carriers may or may not have been treated with an anthracycline-based chemotherapy regimen.
* Approximately at least 12 months from initiation of adjuvant treatment or neo-adjuvant chemotherapy
* Able to provide informed consent

Exclusion Criteria

* Stage IV Breast Cancer
* Genetic testing confirming a variant of unknown significance (VUS) or benign polymorphism in BRCA1 or BRCA2
* V02 Testing contraindicated for any reason, including:

  * Myocardial infarction (within past 3 months)
  * High-risk unstable angina;
  * High-risk or uncontrolled cardiac arrhythmias;
  * Symptomatic severe aortic stenosis;
  * Uncontrolled symptomatic heart failure;
  * Acute pulmonary embolus or pulmonary infarction;
  * Acute myocarditis or pericarditis;
  * Acute aortic dissection;
  * Coronary revascularization procedure within the past three months;
  * Uncontrolled hypertension, defined as systolic blood pressure ≥ 180mmHg or diastolic blood pressure ≥ 100mmHg;
  * Clinically significant valvular heart disease (severe stenosis or regurgitation);
  * Known aortic aneurysm; or
  * Any other condition which, in the opinion of the investigator, may impede testing of the study hypothesis or make it unsafe to engage in the V02 test
* Women who are pregnant
* Any other clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Initial diagnosis of Breast Cancer in 2005 or later BRCA testing documenting either germline mutation in BRCA1/BRCA2 or no mutation in BRCA1/2.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ky, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided